CLINICAL TRIAL: NCT02853526
Title: Transjugular Intrahepatic Portosystemic Shunt (TIPS) for Variceal Rebleeding in Cirrhotic Patients With Occlusive Portal Vein Thrombosis (PVT) and Cavernous Transformation of the Portal Vein (CTPV)
Brief Title: TIPS for Variceal Rebleeding in Cirrhotic Patients With Occlusive Portal Vein Thrombosis and CTPV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zaibo Jiang (Other)
Responsible Party: Sponsor-Investigator, Zaibo Jiang, Head of the intervention and vascular surgery department, the Third Affiliated Hospital, Sun Yat-sen University, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIPSVRDORNO3HSYSU
Record Dates: First submitted 2016-07-24; First posted 2016-08-03 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-07

CONDITIONS: Portal Vein, Cavernous Transformation of; Portal Vein Thrombosis; Liver Cirrhosis; Bleeding Esophageal Varices
MeSH Terms: conditions — Portal Vein, Cavernous Transformation Of; Liver Cirrhosis | interventions — Portasystemic Shunt, Transjugular Intrahepatic; Propranolol; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIPS arm (Experimental): Transjugular intrahepatic portosystemic shunt(TIPS) is an artificial channel within the liver that establishes communication between the inflow portal vein and the outflow hepatic vein. It is used to treat portal hypertension.TIPS was performed in a conventional fashion or in combination of percutaneous transhepatic or transsplenic approach (also called p-TIPS or modified TIPS). Oral warfarin was used for six months to one year prescribed at dosages to achieve an international normalized ratio (INR) of up to two times the upper limit of normal for the prevention of shunt dysfunction.
  Interventions: Procedure: TIPS; Drug: Warfarin
- conservative treatment arm (Active Comparator): Conservative treatment including endoscopic therapy，non-selective beta blockers (propranolol)and anticoagulation therapy (warfarin).
  Interventions: Drug: Propranolol; Procedure: Endoscopic therapy; Drug: Warfarin

INTERVENTIONS:
Procedure: TIPS — Transjugular intrahepatic portosystemic shunt(TIPS)- TIPS was performed in a conventional fashion or in combination of percutaneous transhepatic or transsplenic approach (p-TIPS). Oral warfarin was used for six months to one year prescribed at dosages to achieve an international normalized ratio (INR) of up to two times the upper limit of normal for the prevention of shunt dysfunction.
  Other Names: Transjugular intrahepatic portosystemic shunt
  Arms: TIPS arm
Drug: Propranolol — Propranolol is a kind of non-selective beta blockers, and is used for reducing the portal pressure.
  Arms: conservative treatment arm
Procedure: Endoscopic therapy — Endoscopic therapy includes the endoscopic variceal band ligation and sclerotherapy.
  Arms: conservative treatment arm
Drug: Warfarin — Oral warfarin was used for six months to one year prescribed at dosages to achieve an international normalized ratio (INR) of up to two times the upper limit of normal.

SUMMARY:
To date, there is no treatment strategies for these patients according to American Association of the Study of Liver Disease (AASLD) practice guidelines and Baveno V consensus. Thus, we aim to compare the safety and efficacy of TIPS and conservative treatment (non-selective beta blockers, endoscopic therapy and/or anticoagulation) in patients with PVT and CPTV.

DETAILED DESCRIPTION:
The incidence of portal vein thrombosis (PVT) is about 16% in cirrhotic patients. Chronic PVT often cause two main undesirable consequences: symptomatic portal hypertension (such as variceal bleeding or ascites) and cavernous transformation of portal vein (CPTV). The former could lead to death and the latter increases the difficulty of the transjugular intrahepatic portosystemic shunt (TIPS) treatment, which is considered as a main effective treatment for symptomatic portal hypertension. Some patients with CPTV and variceal bleeding only have to receive conservative treatment (non-selective beta blockers, endoscopic therapy and/or anticoagulation). With advances in technology, modified TIPS procedure could significantly improve the operation success rate of patients with CPTV. To date, the difference in safety and efficacy between TIPS and conservative treatment (non-selective beta blockers, endoscopic therapy and/or anticoagulation) in patients with PVT and CPTV is still unclear.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosis with portal vein thrombosis and cavernous transformation of portal vein and portal hypertension by contrast enhanced CT or MRI.
* History of variceal bleeding.
* Liver cirrhosis.
* Neutrophilous counts≥ 1.5×109/L, Platelet counts ≥ 50 × 109/L, Hemoglobin≥ 85g/L.
* Albumin ≥2.8 g/dL, total bilirubin <51.3 umol/L; alanine aminotransferase (ALT) and aspartate transaminase（AST）<5 times of upper limit.
* PT(Prothrombin time)-INR(international normalized ratio) < 1.7.

Exclusion Criteria:

* Thrombosis involve superior mesenteric vein, splenic vein, or the whole portal vein system. Not suitable for TIPS (judged by principal investigator).
* Company with malignant tumors in liver or other organs.
* Patients with known severe dysfunction of heart, lung, brain or kidney.
* Active bleeding.
* Not eligible for anticoagulation therapy,non-selective beta blockers or endoscopic therapy.
* Uncontrolled infection.
* Pregnancy and breastfeeding.
* HIV infection.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Variceal rebleeding | 3 years
  Variceal rebleeding rate in 3 years

SECONDARY OUTCOMES:
Overall survival time | 3 years
Variceal rebleeding-related death rate | 3 years
Treatment-related complications | 3 years
  Incidence of treatment-related complications
Transjugular intrahepatic portosystemic shunt success rate | 3 years
  Technical success rate of transjugular intrahepatic portosystemic shunt

CONTACTS AND LOCATIONS:
Overall Officials: Zaibo Jiang, Principal Investigator — Department of Intervention and Vascular Surgery, the Third Affiliated Hospital, Sun Yat-sen University
Locations (1):
- Department of Radiology, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided